CLINICAL TRIAL: NCT06590051
Title: AMG 335 Expanded Access Program for IgG4-Related Disease
Status: Available | Type: Expanded Access
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: AMG335 Expanded Access Program
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: UPLIZNA

SUMMARY:
Expanded access requests for AMG 335 may be considered for adult patients with a confirmed diagnosis of IgG4-related disease. To request access, use Responsible Party contact information provided in this record.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen